CLINICAL TRIAL: NCT02894138
Title: Optimal Coronary Flow After PCI for Myocardial Infarction - a Pilot Study
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OPTIMAL-01
Record Dates: First submitted 2016-08-24; First posted 2016-09-09 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: ST-segment Elevation Myocardial Infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Alteplase (Experimental): 40 patients: 4-5 minutes of infusion of 10 ml of alteplase 2mg/ml in culprit vessel
  Interventions: Drug: alteplase
- Placebo (Placebo Comparator): 40 patients: 4-5 minutes of infusion of 10 ml of NaCl in culprit vessel
  Interventions: Drug: Placebo
- Observational (No Intervention): 10 patients with IMR <30 will undergo the same follow-up as the randomised patients

INTERVENTIONS:
Drug: alteplase
  Other Names: Actilyse®
  Arms: Alteplase
Drug: Placebo
  Other Names: NaCl
  Arms: Placebo

SUMMARY:
In this study the investigators test the hypothesis that alteplase given intra coronary after PCI reduce infarct size in patients with ST-elevation myocardial infarction(STEMI) and impaired microvascular function defined as a value of index of microvascular resistance (IMR) >30.

DETAILED DESCRIPTION:
After coronary stenting, index of microvascular resistance (IMR) will be measured invasively. Patients with IMR >30 will be randomised to 20 mg alteplase or placebo (NaCl) administered in the culprit vessel through a microcatheter. Magnet resonance imaging (MRI) of the myocardium will be performed early (2-6 days) and late (3 months) to estimate the primary endpoint (infarct size).

10 non-randomised patients, with IMR <30, will undergo the same follow-up as the randomised patients.

Clinical events for all randomised and non-randomised patients will be collected from Swedish national registries and by telephone at 3 and 12 months.

ELIGIBILITY:
Criteria for randomization:

1. IMR measured in culprit vessel > 30

Criteria for IMR measurement:

Inclusion Criteria:

1. Oral and signed informed consent
2. Males and females 18 - 85 years of age
3. Diagnosis of ST-elevation myocardial infarction (STEMI) including occlusion of culprit vessel on angiography
4. Onset of continuous symptoms within 12 hours
5. Have undergone PCI of culprit vessel
6. Subjects are willing to comply with scheduled visits and tests and are able and willing to provide informed consent

Exclusion Criteria:

1. Previously known ejection fraction <30%
2. Previous PCI in the culprit vessel
3. Chronic total occlusion in major vessel
4. Any history of bleeding diathesis, known coagulopathy, or will refuse blood transfusions
5. Recent history or known platelet count <100.000 cells/mm3 or Hbg < 10 g/dL
6. Known reduced kidney function with estimated glomerular filtration rate (GFR) <30 ml/min/1.73m2.
7. Previous hemorrhagic stroke
8. Ongoing oral anticoagulation treatment
9. Severe asthma requiring daily treatment
10. Any mechanical complication (e.g. ventricular septal defect, papillary muscle rupture, cardiac tamponade)
11. Atrioventricular block grade III
12. Known inability to undergo MRI investigation

    Permanent pacemaker
    * Pronounced claustrophobia
13. Known intolerance to study drug
14. Known intolerance to adenosine
15. Pregnancy
16. Participation in another investigational drug study
17. Previous randomization in the OPTIMAL-PCI trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-09; Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Ratio of myocardial infarct size to area at risk assessed by MRI | 3 months
  MRI performed early (day 2-6) to assess area at risk and late (3 months) to assess infarct size

SECONDARY OUTCOMES:
Change of index of microvascular resistance and coronary flow reserve | Immediately after drug administration during invasive index procedure
  Difference in invasively measured IMR and CFR before and after drug administration
Degree of microvascular obstruction assessed by MRI | 2-6 days
  Degree of microvascular obstruction assessed by MRI
Peak level of Troponin T | 12 hours
  Peak level of Troponin T
Level of NtProBNP | 12 hours
  Level of NtProBNP
Non invasive CFR | 3 months
  CFR measured with transthoracic echo doppler
Major adverse cardiac event (myocardial infarction, stroke, heart failure or death) | 3 months
  Major adverse cardiac event (myocardial infarction, stroke, heart failure or death)
Major adverse cardiac event (myocardial infarction, stroke, heart failure or death) | 12 months
  Major adverse cardiac event (myocardial infarction, stroke, heart failure or death)
Re-hospitalisation for heart failure | 12 months
  Re-hospitalisation for heart failure
Re-hospitalisation for myocardial infarction | 12 months
  Re-hospitalisation for myocardial infarction
Cardiovascular death | 12 months
  Cardiovascular death
Bleeding according to BARC-criteria | 7 days
  Bleeding events during or after index PCI during index hospitalisation
Myocardial hemorrhage at MRI | 2-6 days
  Myocardial hemorrhage at MRI
Change in hemoglobin | 12 hours
  Change in hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Angerås, MD, PhD, Principal Investigator — Department of Cardiology, Sahlgrenska University Hospital, Gothenburg, Sweden
Locations (1):
- Department of Cardiology, Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fearon WF, Shah M, Ng M, Brinton T, Wilson A, Tremmel JA, Schnittger I, Lee DP, Vagelos RH, Fitzgerald PJ, Yock PG, Yeung AC. Predictive value of the index of microcirculatory resistance in patients with ST-segment elevation myocardial infarction. J Am Coll Cardiol. 2008 Feb 5;51(5):560-5. doi: 10.1016/j.jacc.2007.08.062. PMID 18237685
- [Background] Lim HS, Yoon MH, Tahk SJ, Yang HM, Choi BJ, Choi SY, Sheen SS, Hwang GS, Kang SJ, Shin JH. Usefulness of the index of microcirculatory resistance for invasively assessing myocardial viability immediately after primary angioplasty for anterior myocardial infarction. Eur Heart J. 2009 Dec;30(23):2854-60. doi: 10.1093/eurheartj/ehp313. Epub 2009 Aug 14. PMID 19684025
- [Background] Fearon WF, Low AF, Yong AS, McGeoch R, Berry C, Shah MG, Ho MY, Kim HS, Loh JP, Oldroyd KG. Prognostic value of the Index of Microcirculatory Resistance measured after primary percutaneous coronary intervention. Circulation. 2013 Jun 18;127(24):2436-41. doi: 10.1161/CIRCULATIONAHA.112.000298. Epub 2013 May 16. PMID 23681066
- [Background] Boscarelli D, Vaquerizo B, Miranda-Guardiola F, Arzamendi D, Tizon H, Sierra G, Delgado G, Fantuzzi A, Estrada D, Garcia-Picart J, Cinca J, Serra A. Intracoronary thrombolysis in patients with ST-segment elevation myocardial infarction presenting with massive intraluminal thrombus and failed aspiration. Eur Heart J Acute Cardiovasc Care. 2014 Sep;3(3):229-36. doi: 10.1177/2048872614527008. Epub 2014 Mar 17. PMID 24637066
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242